CLINICAL TRIAL: NCT02463422
Title: Detection of ASD at the 1st Birthday as Standard of Care: The Get SET Early Model
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: Southwest Autism Research and Resource Center (SARRC) (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karen Pierce, Co-Director of the Autism Center of Excellence, University of California, San Diego
Other Study IDs: R01MH104446 (NIH); R01MH104446 (NIH)
Record Dates: First submitted 2015-05-27; First posted 2015-06-04 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- San Diego, CA: Toddlers detected with ASD and other disorders based on the Get SET Early Model in San Diego.
- Phoenix, AZ: Toddlers detected with ASD and other disorders based on the Get SET Early Model in Phoenix.

SUMMARY:
According to a recent report from the Centers for Disease Control, most children with ASD do not receive a diagnosis and begin receiving treatment until well after their 4th birthday, which is unfortunate given that many connections between brain cells have already been established by that age. This program will test a model called Get S.E.T. Early (S=Screen, E=Evaluate, T=Treat) in both San Diego and Phoenix, designed to detect, evaluate, and treat ASD within the first 2 years of life. In this proposal 7,500 toddlers from the general population will be screened in San Diego and Phoenix (total 15,000) using the CSBS IT Checklist (Wetherby & Prizant, 2002) at well baby check-ups using a "triple screen" approach wherein toddlers are screened at three ages starting at 12 months. Investigators predict that providing screening tools with clear cut-off scores and guidelines for automatic referral for both evaluation and treatment will result in dramatically lowering mean age of detection in Phoenix from 4-5 years down to 1-2 years. Investigators also predict that using repeat screening at 12, 18, & 24 months in combination with automatic referral options via technology (i-Pads) will result in an increase in the number of ASD toddlers detected by 24 months relative to a single time point screen using traditional paper screens.

DETAILED DESCRIPTION:
Investigators previously demonstrated that their early intervention model system, which was centered on using the CSBS IT Checklist to screen all babies at the 1-year check-up as standard of care, resulted in a mean age of 12 months for screening, 14 months for evaluation, and 18 months for treatment participation. These are far younger ages than is common in the U.S. The 3-stage model system, Get SET (S=Screen; E=Evaluate; T=Treat) Early, screened >10,000 1 year olds in the first trial run detecting over 100 ASD and other developmental delayed toddlers. The current grant will build on this highly effective model by implementing a new version in two major cities: San Diego and Phoenix; data mined from electronic records from Kaiser pediatric offices in Los Angeles and Irvine will provide control data. In Phoenix, investigators test the feasibility of establishing the Get SET Early model in a city with one of the lowest median incomes and oldest age of first diagnosis in America. In AIM #1, the Screen and Refer Early stage, investigators will create a Pediatrician Network with 100 members in Phoenix. In San Diego investigators will utilize their existing Pediatrician Network and test new innovations such as a repeat "triple screen" at 12, 18, and 24 months to ensure that no toddlers are missed. Speed of referral for evaluation will be compared and contrasted using parent (self) and automatic (referral i-Pad App) options. Investigators will track every toddler with an eventual ASD diagnosis within circumscribed medical groups to determine the true sensitivity and specificity of the screening tool and the percentage of ASD toddlers detected by this model. Anonymous survey data regarding screening habits will be administered to parents and pediatricians. AIM #2 implements the Evaluate and Refer Early stage. Its key attribute is an ASD Early Evaluation Clinic that specializes in the rapid scheduling and evaluation of every referred screened positive toddler. Toddlers will enter the program at the age they fail the screen (i.e., 12, 18 or 24 months) and will be thoroughly diagnostically evaluated and tracked once per year until they turn 3 years. This specialty Clinic is at the Autism Center in San Diego and will be developed at SARRC in Phoenix. Automated versus optional self-referral for treatment will be tested and compared. AIM #3 implements the Treat Early stage. Its key attributes are a network of providers of empirically based treatment and the innovative use of an inexpensive and readily available web-based treatment tracking system to document engagement. Treatment Networks will be created in San Diego and Phoenix. Primary outcome measures include rates and ages of screening and referral, evaluation and referral, and treatment engagement; sustainability across years; diagnostic, clinical and demographic characteristics of subjects; professional and parent satisfaction at each stage. Investigators hypothesize that providing screening tools with clear cut-off scores and guidelines for automatic referral for evaluation and treatment, will result in dramatically lowering mean age of diagnosis and treatment in Phoenix from 4-5 years down to 1-2 years; San Diego will likewise have mean ages of 1-2 years for diagnosis and treatment making them significantly earlier than non-intervention contrast cities.

ELIGIBILITY:
Inclusion Criteria:

* Completed CSBS IT Checklist at pediatrician office
* Pediatrician referred
* Between 12 and 36 months

Exclusion Criteria:

* Older than 36 months

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Two cohorts of toddlers, those in San Diego and Phoenix, will participate. Toddlers in both cities from the general population will be screened for ASD and other delays using the CSBS Infant-Toddler Checklist in pediatric offices at the 12, 18, and 24 month well-baby visits.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Rate of screening per pediatric office | Year 4
Rate of referral for developmental evaluation per pediatric office | Year 4
Age at screen | Year 4
Age at developmental evaluation | Year 4
Age at treatment start | Age at treatment start will be tracked for 4 years, and an average age computed in year 5
Number of ASD toddlers detected by program | Year 4
Changes in parent and pediatrician screening perceptions from baseline to Year 4 | Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Karen Pierce, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Southwest Autism Research & Resource Center (Sarrc), Phoenix, Arizona
  - Autism Center of Excellence, La Jolla, California